CLINICAL TRIAL: NCT00003551
Title: A Phase II Study of 9-Amino-20(S)-Camptothecin (9-AC) (NSC 603071) and Evaluation of Drug Resistance in Patients With Advanced Renal Cell Carcinoma
Brief Title: Aminocamptothecin in Treating Patients With Advanced or Recurrent Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066608; EUSM-HIC-748-96; NCI-T96-0110
Record Dates: First submitted 1999-11-01; First posted 2004-09-13 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2000-07

CONDITIONS: Kidney Cancer
Keywords: stage III renal cell cancer; stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell

INTERVENTIONS:
Drug: aminocamptothecin colloidal dispersion

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of aminocamptothecin in treating patients with stage III, stage IV, or recurrent kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate, duration of response, and survival of patients with advanced renal cell carcinoma treated with aminocamptothecin colloidal dispersion. II. Determine the nature and degree of toxicity of aminocamptothecin in this patient population.

OUTLINE: Patients receive aminocamptothecin colloidal dispersion intravenously for 120 hours weekly for 2 weeks followed by 1 week of rest. Courses are repeated every 3 weeks in the absence of disease progression or dose limiting toxicity. Patients are followed every 3 months for the first 2 years, every 6 months for the next 3 years, and yearly thereafter.

PROJECTED ACCRUAL: A total of 10-29 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven stage III, stage IV, or recurrent renal cell carcinoma Measurable disease No brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: Platelet count at least 100,000/mm3 Absolute neutrophil count at least 1500/mm3 Hemoglobin at least 9.0 g/dL Hepatic: Bilirubin no greater than 1.5 mg/dL ALT and AST no greater than 2.5 times the institutional normal values Renal: Creatinine no greater than 1.5 mg/dL Other: Not pregnant or nursing Fertile patients must use effective contraception No uncontrolled systemic infection No other prior or concurrent malignancies except nonmelanoma skin cancer, carcinoma in situ of the cervix, or ductal carcinoma in situ of the breast that have been curatively treated No evidence of delirium, confusion, suicidal ideation, or untreated depression

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 30 days since prior cytokines and recovered No more than 1 prior treatment with cytokines (interleukin-2 or interferons) Chemotherapy: No prior cytotoxic chemotherapy No prior aminocamptothecin No other concurrent antineoplastic agents Endocrine therapy: At least 30 days since prior hormone therapy and recovered No more than 1 prior hormone therapy (tamoxifen or medroxyprogesterone) Radiotherapy: Prior radiotherapy allowed if indicator lesion and greater than 15% of marrow producing bone have not been irradiated Surgery: Recovered from prior surgery Other: At least 30 days since other investigational agents No concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-08; Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Keane, MD, Study Chair — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Emory University School of Medicine, Atlanta, Georgia